CLINICAL TRIAL: NCT01898494
Title: Phase II Randomized Trial of Transoral Surgical Resection Followed by Low-Dose or Standard-Dose IMRT in Resectable p16+ Locally Advanced Oropharynx Cancer
Brief Title: Transoral Surgery Followed By Low-Dose or Standard-Dose Radiation Therapy With or Without Chemotherapy in Treating Patients With HPV Positive Stage III-IVA Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3311; NCI-2013-00814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E3311 (Other: ECOG-ACRIN Cancer Research Group); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Human Papilloma Virus Infection; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Oropharynx
Keywords: oropharynx cancer; HPV+
MeSH Terms: conditions — Papillomavirus Infections; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Platinum; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm S (Surgery) then Arm A (Low risk, observation) (Experimental): Patients undergo transoral surgical resection of the oropharyngeal tumor. After transoral surgical resection of the oropharyngeal tumor, low risk patients are under observation.
  Interventions: Procedure: Transoral surgery
- Arm S (Surgery) then Arm B (Intermediate risk, low-dose IMRT) (Experimental): Patients undergo transoral surgical resection of the oropharyngeal tumor. After transoral surgical resection of the oropharyngeal tumor, intermediate risk patients receive low-dose IMRT (50 Gy) QD five days a week for 5 weeks.
  Interventions: Procedure: Transoral surgery; Radiation: intensity-modulated radiation therapy
- Arm S (Surgery) then Arm C (Intermediate risk, standard-dose IMRT) (Experimental): Patients undergo transoral surgical resection of the oropharyngeal tumor. After transoral surgical resection of the oropharyngeal tumor, intermediate risk patients receive standard-dose IMRT (60 Gy) QD five days a week for 6 weeks.
  Interventions: Procedure: Transoral surgery; Radiation: intensity-modulated radiation therapy
- Arm S (Surgery) then Arm D (High risk, IMRT, chemotherapy) (Experimental): Patients undergo transoral surgical resection of the oropharyngeal tumor. After transoral surgical resection of the oropharyngeal tumor, high risk patients then receive IMRT (66Gy) QD five days a week for 6-7 weeks. Patients also receive cisplatin IV over 60 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiation therapy.
  Interventions: Procedure: Transoral surgery; Radiation: intensity-modulated radiation therapy; Drug: cisplatin; Drug: carboplatin

INTERVENTIONS:
Procedure: Transoral surgery — Undergo transoral surgical resection
  Other Names: TOS
Radiation: intensity-modulated radiation therapy — Undergo standard-dose or low-dose IMRT
  Other Names: IMRT
  Arms: Arm S (Surgery) then Arm B (Intermediate risk, low-dose IMRT); Arm S (Surgery) then Arm C (Intermediate risk, standard-dose IMRT); Arm S (Surgery) then Arm D (High risk, IMRT, chemotherapy)
Drug: cisplatin — Given IV
  Other Names: Cis-diaminedichloroplatinum Cis-diaminedichloroplatinum (II); diaminedichloroplatinum; cis-platinum; CDDP; DDP; platinum; Platinol; Platinol-AQ; DACP; NSC 119875 R R
  Arms: Arm S (Surgery) then Arm D (High risk, IMRT, chemotherapy)
Drug: carboplatin — Given IV
  Other Names: CBDCA; JM-8; NSC-241240; Paraplatin
  Arms: Arm S (Surgery) then Arm D (High risk, IMRT, chemotherapy)

SUMMARY:
This randomized phase II trial studies how well transoral surgery followed by low-dose or standard-dose radiation therapy works in treating patients with human papilloma virus (HPV) positive stage III-IVA oropharyngeal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy with chemotherapy may kill any tumor cells that remain after surgery. It is not yet known how much extra treatment needs to be given after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Accrual, risk distribution, and surgical quality will be used to determine the feasibility of a prospective multi-institutional study of transoral surgery for HPV positive (+) oropharynx cancer followed by risk-adjusted adjuvant therapy.

II. To assess the oncologic efficacy following transoral resection and adjuvant therapy in patients determined to be at "intermediate risk" after surgical excision, the 2-year progression free survival (PFS) rate will be examined.

SECONDARY OBJECTIVES:

I. To estimate the patient distribution with various histologic risk features. II. To assess and compare early and late toxicities associated with transoral surgery (TOS) and the different doses of adjuvant postoperative radiotherapy (PORT).

III. To evaluate swallowing function before and after TOS and risk-adjusted adjuvant therapy.

IV. To evaluate quality of life (QOL), swallowing perception and performance, voice outcomes, and head and neck symptoms.

TERTIARY OBJECTIVES:

I. To correlate tumor TP53 mutation and other associated mutation profile with pathologic findings, with PFS and other outcome parameters in patients with resectable HPV-associated oropharyngeal squamous cell carcinoma (OPSCC) after the above treatments.

II. To evaluate radiation resistance markers, including excision repair cross complementing 1 (ERCC1) single nucleotide polymorphism and protein expression, and correlate them with treatment efficacy.

III. To investigate the usefulness of biomarkers in predicting progression-free survival and biomarkers, including tumor ERCC1, epidermal growth factor receptor (EGFR), plasma cytokine/chemokines, cellular immunity to HPV, and oral HPV deoxyribonucleic acid (DNA).

OUTLINE: All patients undergo transoral surgery (TOS) in Step 1.

ARM S: Patients undergo transoral resection of the oropharyngeal tumor.

Then patients are classified by risk status (low risk, intermediate risk, or high risk) in Step 2 and assigned to the appropriate treatment group. Patients classified as intermediate risk are randomized to arms B or C.

ARM A (low risk; observation): Patients receive observation.

ARM B (intermediate risk): Patients undergo low-dose (50Gy) intensity modulated radiation therapy (IMRT) once daily (QD) over 25 fractions.

ARM C (intermediate risk): Patients undergo standard-dose (60Gy) IMRT QD over 30 fractions.

ARM D (high risk): Patients receive IMRT at 66 Gy QD for 33 fractions. Patients also receive cisplatin intravenously (IV) over 60 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiation therapy.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 year.

ELIGIBILITY:
Inclusion Criteria:

Registration to Surgery (Arm S)

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have newly diagnosed, histologically or cytologically confirmed squamous cell carcinoma or undifferentiated carcinoma of the oropharynx; patients must have been determined to have resectable oropharyngeal disease; patients with primary tumor or nodal metastasis fixed to the carotid artery, skull base or cervical spine are not eligible
* Patients must have American Joint Committee on Cancer (AJCC) TNM tumor stage III, IV a, or IV b (with no evidence of distant metastases) as determined by imaging studies (performed < 30 days prior to pre-registration) and complete head and neck exam; the following imaging is required: computed tomography (CT) scan with IV contrast or magnetic resonance imaging (MRI)
* Patients must have biopsy-proven p16+ oropharynx cancer; the histologic evidence of invasive squamous cell carcinoma may have been obtained from the primary tumor or metastatic lymph node. It is required that patients have a positive p16 IHC (as surrogate for HPV) status from either the primary tumor or metastatic lymph node.
* Carcinoma of the oropharynx associated with HPV as determined by p16 protein expression using immunohistochemistry (IHC) performed by a Clinical Laboratory Improvement Amendments (CLIA) approved laboratory; using p16 antibody obtained from Roche mtm laboratories AG (CINtec, clone E6H4) is recommended
* Patients with a history of a curatively treated malignancy must be disease-free for at least two years except for carcinoma in situ of cervix and/or non-melanomatous skin cancer
* Patients with the following within the last 6 months prior to pre-registration must be evaluated by a cardiologist and/or neurologist prior to entry into the study

  * Congestive heart failure > NYHA Class II
  * Cerebrovascular accident (CVA)/transient ischaemic attack (TIA)
  * Unstable angina
  * Myocardial infarction
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< the upper limit of normal (ULN)
* Calculated creatinine clearance must be > 60 ml/min using the Cockcroft-Gault formula

Registration/Randomization to Step2 - Arms A, B, C and D

* Histopathologic assessment of surgical pathology must include examination for perineural invasion (PNI) and lymphovascular invasion (LVI) and reported as absent or present; the absence or presence of extracapsular extension (ECE) requires gross and microscopic assessment and is defined to be:

  * Absent (negative or nodal metastasis with smooth/rounded leading edge confined to thickened capsule/pseudocapsule),
  * Present - minimal (tumor extends =< 1 mm beyond the lymph node capsule), or
  * Present - extensive (gross, tumor extends > 1 mm beyond the lymph node capsule (includes soft tissue metastasis)
* Patient must be stratified/classified into one of the following risk categories (the highest risk feature assessed pathologically will determine the patient's category/treatment arm assignment):

  * Low Risk: T1-T2, N0-N1 AND clear (≥ 3mm) margins, AND no ECE or PNI/LVI
  * High Risk: Any of the following features: one or more positive margin(s) with any T stage, OR "Extensive" (> 1mm) ECE, OR ≥ 5 metastatic lymph nodes (regardless of primary tumor margin status)
  * Intermediate Risk: Any of the following features: one or more "close" (< 3mm) margin(s), OR "Minimal" (≤ 1mm) ECE, OR N2a (1 or more lymph node > 3cm in diameter), OR N2b (2-4 lymph nodes positive, any diameter ≤ 6cm), OR with perineural invasion or lymphovascular invasion.
  * Unknown Risk: Patients found to have N2C or N3 disease on final pathologic analysis are at unknown risk for recurrence, but are not candidates for deintensified adjuvant therapy in this trial. These patients will be treated on Arm C.
  * Patients not categorized into the appropriate risk category will be considered ineligible for the study
* Patient must be registered/randomized to Step 2 within a maximum of 7 weeks following surgery
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception

Exclusion Criteria:

Registration to Surgery (Arm S)

* Prior radiation above the clavicles
* Evidence of extensive or "matted/fixed" pathologic adenopathy on preoperative imaging
* Women must not be pregnant or breast-feeding due to the teratogenicity of chemotherapy; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Any intercurrent illness likely to interfere with protocol therapy or prevent surgical resection
* Uncontrolled diabetes, uncontrolled infection despite antibiotics or uncontrolled hypertension within 30 days prior to pre-registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ferris, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (58):
- United States (58):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Stanford Cancer Institute, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Miami Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mercy Hospital Springfield, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Hospitals, Norfolk, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Ferris RL, Flamand Y, Weinstein GS, Li S, Quon H, Mehra R, Garcia JJ, Chung CH, Gillison ML, Duvvuri U, O'Malley BW Jr, Ozer E, Thomas GR, Koch WM, Gross ND, Bell RB, Saba NF, Lango M, Mendez E, Burtness B. Phase II Randomized Trial of Transoral Surgery and Low-Dose Intensity Modulated Radiation Therapy in Resectable p16+ Locally Advanced Oropharynx Cancer: An ECOG-ACRIN Cancer Research Group Trial (E3311). J Clin Oncol. 2022 Jan 10;40(2):138-149. doi: 10.1200/JCO.21.01752. Epub 2021 Oct 26. PMID 34699271
- [Derived] Burtness B, Flamand Y, Quon H, Weinstein GS, Mehra R, Garcia JJ, Kim S, O'Malley BW Jr, Ozer E, Ikpeazu C, Koch WM, Gross ND, Bell RB, Patel M, Lango MN, Morris LG, Smith R, Karakla D, Richmon JD, Holsinger FC, Ferris RL. Long-Term Follow-Up of E3311, an ECOG-ACRIN Cancer Research Group Phase II Trial of Transoral Surgery and Risk-Based Adjuvant Treatment in Human Papillomavirus-Initiated Oropharynx Cancer. J Clin Oncol. 2025 Aug 10;43(23):2559-2565. doi: 10.1200/JCO-24-02550. Epub 2025 Jun 10. PMID 40493877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on July 9, 2013, accrued its first patient on January 22, 2014, and closed to accrual on July 7, 2017 for a total of 519 patients.
Groups:
- Arm S (Transoral Surgery) Then Arm A (Observation): Patients receive observation after transoral surgery.
- Arm S (Transoral Surgery) Then Arm B (Radiotherapy IMRT 50 Gy): Patients under go transoral surgery and then receive low-dose (50Gy) intensity modulated radiation therapy (IMRT) once daily (QD) over 25 fractions.
- Arm S (Transoral Surgery) Then Arm C (Radiotherapy IMRT 60 Gy): Patients undergo transoral surgery and then receive standard-dose (60Gy) IMRT QD over 30 fractions.
- Arm S (Transoral Surgery) Then Arm D (Chemo + IMRT 66 Gy): Patients undergo transoral surgery and then receive IMRT at 66 Gy QD for 33 fractions. Patients also receive cisplatin intravenously (IV) over 60 minutes or carboplatin IV over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiation therapy.
- Not Being Assigned to Step 2 Adjuvant Treatment Arms: Patients either did not receive transoral surgery at Step 1 or were not assigned to Step 2 treatment arms.
Period: Step 1 (Arm S - Transoral Surgery)
Arm/Group | Arm S (Transoral Surgery) Then Arm A (Observation) | Arm S (Transoral Surgery) Then Arm B (Radiotherapy IMRT 50 Gy) | Arm S (Transoral Surgery) Then Arm C (Radiotherapy IMRT 60 Gy) | Arm S (Transoral Surgery) Then Arm D (Chemo + IMRT 66 Gy) | Not Being Assigned to Step 2 Adjuvant Treatment Arms
Started | 49 | 126 | 132 | 138 | 74
Completed | 49 | 126 | 132 | 138 | 50
Not Completed | 0 | 0 | 0 | 0 | 24
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Patient ineligible | 0 | 0 | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 9
Not completed — Disease progression | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Alternative therapy | 0 | 0 | 0 | 0 | 1
Not completed — Surgery planned but not performed | 0 | 0 | 0 | 0 | 1
Period: Step 2 (Adjuvant Treatment)
Arm/Group | Arm S (Transoral Surgery) Then Arm A (Observation) | Arm S (Transoral Surgery) Then Arm B (Radiotherapy IMRT 50 Gy) | Arm S (Transoral Surgery) Then Arm C (Radiotherapy IMRT 60 Gy) | Arm S (Transoral Surgery) Then Arm D (Chemo + IMRT 66 Gy) | Not Being Assigned to Step 2 Adjuvant Treatment Arms
Started | 49 | 126 | 132 | 138 | 0 (This group of patients did not proceed to adjuvant treatment on this study. They either received surgery but did not proceed to adjuvant treatment or did not receive surgery in Step 1.)
Treated | 49 | 120 | 127 | 134 | 0
Eligible and Treated | 38 | 100 | 108 | 113 | 0
Eligible and Treated Patients With Baseline MDADI Assessed | 35 | 91 | 99 | 102 | 0
Eligible and Treated Patients With Post-surgery MDADI Assessed | 31 | 83 | 88 | 94 | 0
Eligible and Treated Patients With FACT-H&N Assessed at 6 Months | 21 | 75 | 80 | 77 | 0
Completed | 49 | 119 | 118 | 127 | 0
Not Completed | 0 | 7 | 14 | 11 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Alternative therapy | 0 | 0 | 1 | 0 | 0
Not completed — Never started treatment | 0 | 6 | 5 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Arm S (Surgery) Then Arm D (High Risk, IMRT, Chemotherapy): Patients undergo transoral surgical resection of the oropharyngeal tumor. After transoral surgical resection of the oropharyngeal tumor, high risk patients then receive IMRT (66Gy) QD five days a week for 6-7 weeks. Patients also receive cisplatin IV over 60 minutes or carboplatin over 30 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiation therapy.
  Transoral surgery: Undergo transoral surgical resection
  intensity-modulated radiation therapy: Undergo standard-dose or low-dose IMRT
  cisplatin: Given IV
  carboplatin: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm S (Surgery) Then Arm A (Low Risk, Observation) | Arm S (Surgery) Then Arm B (Intermediate Risk, Low-dose IMRT) | Arm S (Surgery) Then Arm C (Intermediate Risk, Standard-dose IMRT) | Arm S (Surgery) Then Arm D (High Risk, IMRT, Chemotherapy) | Total
Number analyzed (Participants) | 38 | 100 | 108 | 113 | 359
Age, Continuous [Median (Full Range); unit: years] | 61 [46 to 76] | 59 [42 to 75] | 57 [40 to 77] | 58 [37 to 80] | 58 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 16 | 11 | 40
  Male | 30 | 95 | 92 | 102 | 319
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 4 | 11
  Not Hispanic or Latino | 36 | 90 | 98 | 100 | 324
  Unknown or Not Reported | 0 | 8 | 7 | 9 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 3 | 2 | 9
  White | 35 | 93 | 97 | 106 | 331
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 7 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 2 Years
Description: Progression-free survival is defined as the time from randomization/assignment of post-surgical treatment to the appearance of lesions, including primary, nodal or new site, or death, whichever occurs first. These patients are considered disease-free after surgery so the appearance of any lesions is counted as progression. Kaplan-Meier estimate was used to characterize progression-free survival rate at 2 years.
Time Frame: Assessed every 3 months for 2 years
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm S (Surgery) Then Arm A (Low Risk, Observation) | Arm S (Surgery) Then Arm B (Intermediate Risk, Low-dose IMRT) | Arm S (Surgery) Then Arm C (Intermediate Risk, Standard-dose IMRT) | Arm S (Surgery) Then Arm D (High Risk, IMRT, Chemotherapy)
Number analyzed (Participants) | 38 | 100 | 108 | 113
proportion of participants | 0.969 [0.919 to 1.00] | 0.949 [0.913 to 0.986] | 0.96 [0.928 to 0.993] | 0.907 [0.862 to 0.954]

2. Primary Outcome: Proportion of Patients With Grade III or IV Oropharyngeal Bleeding or Positive Margins
Description: Surgery quality was evaluated based on grade 3-4 bleeding events per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 during surgery and positive margins after surgery. Per CTCAE v5.0, grade 3 = severe and grade 4 = life-threatening.
  Having grade 3-4 bleeding or positive margins indicates worse outcomes.
Time Frame: Assessed during surgery and directly after surgery
Population: Patients who received surgery
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Arm S (Surgery): Patients undergo transoral surgical resection of the oropharyngeal tumor.
Arm/Group | Arm S (Surgery)
Number analyzed (Participants) | 495
proportion of participants | 0.091 [0.071 to 0.115]

3. Secondary Outcome: Distribution of Histologic Risk Status
Description: Low Risk: T1-T2, N0-N1 AND clear (> 3mm) margins, AND no extranodal extension (ENE) or PNI/LVI.
  Intermediate Risk: Any of the following features: one or more "close" (< 3mm) margin(s), OR "Minimal" (< 1mm) ENE, OR N2a (1 or more lymph node >3cm in diameter), OR N2b (2-4 lymph nodes positive, any diameter < 6cm), OR with perineural invastion or lymphovascular invasion.
  High Risk: Any of the following features: one or more positive margin(s) with any T stage, OR "Extensive" (> 1mm) ENE, OR > 5 metastatic lymph nodes (regardless of primary tumor margin status).
Time Frame: Assessed after directly surgery
Population: Patients who received surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm S (Surgery)
Number analyzed (Participants) | 359
Participants
  Low Risk | 38
  Intermediate Risk | 208
  High Risk | 113

4. Secondary Outcome: Swallowing Function Before Surgery Assessed Using MD Anderson Dysphagia Inventory (MDADI)
Description: The MDADI measures swallowing-related quality of life (QOL) in patients with swallowing dysfunction in a 20-item written questionnaire. It evaluates the patient's physical (P), emotional (E) and functional (F) perceptions of swallowing dysfunction. This instrument has been psychometrically validated in head and neck cancer patients. Two summary scores can be obtained from the MDADI: 1) global and 2) composite. The global scale is a single question, scored individually, to assess the overall impact that swallowing abilities have on quality of life ("my swallowing impacts my day-to-day life"). The composite MDADI score summarizes overall performance on remaining 19-items of the MDADI, as a weighted average of the physical, emotional, and functional subscale questions. This study reports the composite MDADI score. The summary MDADI scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning).
Time Frame: Assessed at baseline
Population: Eligible and treated patients with baseline MDADI scores available
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm S (Surgery) Then Arm A (Low Risk, Observation) | Arm S (Surgery) Then Arm B (Intermediate Risk, Low-dose IMRT) | Arm S (Surgery) Then Arm C (Intermediate Risk, Standard-dose IMRT) | Arm S (Surgery) Then Arm D (High Risk, IMRT, Chemotherapy)
Number analyzed (Participants) | 35 | 91 | 99 | 102
score on a scale | 89.1 [84.7 to 93.5] | 90.2 [87.8 to 92.5] | 87.4 [84.6 to 90.1] | 88.2 [85.4 to 91.0]

5. Secondary Outcome: Swallowing Function After Surgery Assessed Using MD Anderson Dysphagia Inventory (MDADI)
Description: as for outcome 4
Time Frame: Assessed 4-6 weeks after surgery
Population: Eligible and treated patients with MDADI scores after surgery available
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm S (Surgery) Then Arm A (Low Risk, Observation) | Arm S (Surgery) Then Arm B (Intermediate Risk, Low-dose IMRT) | Arm S (Surgery) Then Arm C (Intermediate Risk, Standard-dose IMRT) | Arm S (Surgery) Then Arm D (High Risk, IMRT, Chemotherapy)
Number analyzed (Participants) | 31 | 83 | 88 | 94
score on a scale | 75.5 [66.0 to 85.0] | 76.3 [72.4 to 80.1] | 69.6 [65.1 to 74.1] | 73.3 [68.2 to 78.4]

6. Secondary Outcome: Quality of Life (QOL) at 6 Months After Treatment Assessed by Functional Assessment of Cancer Therapy - Head and Neck Cancer (FACT-HN) Total Score
Description: The FACT-H&N (version 4) consists of a cancer-specific questionnaire, FACT-G, in addition to 12 H&N cancer-specific items (the HN subscale). FACT-G is a 27-item measure that assesses general cancer quality of life. FACT-HN total score ranges between 0 and 148. The higher the score, the better the QOL.
Time Frame: Assessed at 6 months after treatment
Population: Eligible and treated patients with FACT-HN total scores 6 months after treatment available
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm S (Surgery) Then Arm A (Low Risk, Observation) | Arm S (Surgery) Then Arm B (Intermediate Risk, Low-dose IMRT) | Arm S (Surgery) Then Arm C (Intermediate Risk, Standard-dose IMRT) | Arm S (Surgery) Then Arm D (High Risk, IMRT, Chemotherapy)
Number analyzed (Participants) | 21 | 75 | 80 | 77
score on a scale | 128.5 [122.1 to 134.9] | 121.02 [116.5 to 125.5] | 117.8 [113.8 to 121.7] | 114.6 [109.3 to 119.9]

7. Other Pre Specified Outcome: Association Between TP53 Mutation and Progression-free Survival
Description: Progression-free survival is defined as the time from registration to the appearance of new metastatic lesions or objective tumor progression or death, whichever occurs first. Kaplan-Meier estimate was used to characterize progression-free survival.
Time Frame: Assessed every 3 months for 2 years, then every 6 months, up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Association Between Radiation Resistance Markers and Progression-free Survival
Description: as for outcome 7
Time Frame: Assessed every 3 months for 2 year, then every 6 months, up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Usefulness of Biomarkers in Predicting Progression-free Survival
Description: as for outcome 7
Time Frame: Assessed every 3 months for 2 years, then every 6 months, up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed weekly during the 7 weeks of treatment, then every 2 months up to 2 years post-registration, then every 6 months up to 3 years post-registration
Description: Serious adverse events are defined as grade 3 or higher adverse events that are possibly, probably, or definitely related to protocol therapy. Other adverse events are defined as grade 1 or grade 2 adverse events that are possibly, probably, or definitely related to protocol therapy with a frequency of at least 5% in a given arm.
  All patients enrolled are included in all-cause mortality analysis. Patients who received treatment with adverse event data available are included in AE analysis.
Groups:
- Arm S (Transoral Surgery): Patients receive transoral surgery.
- Arm A (Observation): Patients receive observation after transoral surgery.
- Arm B (Radiotherapy IMRT 50 Gy): Patients with intermediate risk undergo low-dose (50Gy) intensity modulated radiation therapy (IMRT) once daily (QD) over 25 fractions.
- Arm C (Radiotherapy IMRT 60 Gy): Patients with intermediate risk undergo standard-dose (60Gy) IMRT QD over 30 fractions.
- Arm D (Cisplatin + IMRT 66 Gy): High risk patients receive IMRT at 66 Gy QD for 33 fractions. Patients also receive cisplatin intravenously (IV) over 60 minutes on days 1, 8, 15, 22, 29, 36, and 43 during radiation therapy.
Arm/Group | Arm S (Transoral Surgery) | Arm A (Observation) | Arm B (Radiotherapy IMRT 50 Gy) | Arm C (Radiotherapy IMRT 60 Gy) | Arm D (Cisplatin + IMRT 66 Gy)
All-Cause Mortality (participants affected / at risk) | 24/519 | 1/49 | 4/126 | 7/132 | 9/138
Serious Adverse Events (participants affected / at risk) | 85/495 | 0/49 | 17/120 | 31/127 | 81/134
Other Adverse Events (participants affected / at risk) | 110/495 | 1/49 | 57/120 | 71/127 | 96/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm S (Transoral Surgery) (N=495) | Arm A (Observation) (N=49) | Arm B (Radiotherapy IMRT 50 Gy) (N=120) | Arm C (Radiotherapy IMRT 60 Gy) (N=127) | Arm D (Cisplatin + IMRT 66 Gy) (N=134)
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 6
Hemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 3
Fever (General disorders) | 0 | 0 | 0 | 0 | 1
Neck edema (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 3 | 0 | 0 | 1 | 1
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 31 | 0 | 4 | 6 | 21
Esophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Esophageal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 6 | 14 | 27
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 3 | 10
Oral hemorrhage (Gastrointestinal disorders) | 16 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 4 | 0 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 8 | 9
Intraoperative arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 3 | 25
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 23
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 3
Weight loss (Investigations) | 0 | 0 | 1 | 2 | 9
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 22
Investigations - Other, specify (Investigations) | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dysphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 2 | 5
Respiratory, thoracic and mediastinal disorders - Other, spe (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 5 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm S (Transoral Surgery) (N=495) | Arm A (Observation) (N=49) | Arm B (Radiotherapy IMRT 50 Gy) (N=120) | Arm C (Radiotherapy IMRT 60 Gy) (N=127) | Arm D (Cisplatin + IMRT 66 Gy) (N=134)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 9
Fatigue (General disorders) | 0 | 0 | 3 | 17 | 31
Pain (General disorders) | 27 | 0 | 4 | 4 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 13 | 27 | 19
Dysphagia (Gastrointestinal disorders) | 72 | 1 | 14 | 21 | 30
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 26 | 35 | 43
Nausea (Gastrointestinal disorders) | 0 | 0 | 7 | 6 | 24
Oral pain (Gastrointestinal disorders) | 36 | 0 | 7 | 13 | 19
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 7
Mucosal infection (Infections and infestations) | 0 | 0 | 2 | 6 | 10
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 13 | 32 | 42
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 9
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 10
Weight loss (Investigations) | 0 | 0 | 12 | 19 | 34
White blood cell decreased (Investigations) | 0 | 0 | 1 | 0 | 17
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 9 | 10 | 16
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 10
Dysgeusia (Nervous system disorders) | 0 | 0 | 26 | 32 | 34
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT01898494/Prot_SAP_000.pdf